CLINICAL TRIAL: NCT01767935
Title: A Pilot Study of The Tandem Treatment of Painful Osseous Metastases With Cryoablation Followed by Radiation Therapy
Brief Title: Cryosurgery and Radiation Therapy in Treating Patients With Painful Bone Metastases
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Slow Accruals
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Endocare, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00020528; NCI-2012-02087 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); P30CA012197 (NIH); CCCWFU 97212 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2013-01-11; First posted 2013-01-15 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Bone Metastases; Pain
MeSH Terms: conditions — Pain | interventions — Cryosurgery; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Treatment (cryosurgery and radiation therapy) (Experimental): Patients undergo cryosurgery. Beginning 2 weeks later, patients undergo 1, 10, or 15 fractions of radiation therapy 5 days per week for 1-3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.
  Interventions: Procedure: cryosurgery; Radiation: radiation therapy; Procedure: quality-of-life assessment

INTERVENTIONS:
Procedure: cryosurgery — Undergo cryosurgery
  Other Names: cryoablation; cryosurgical ablation
Radiation: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Procedure: quality-of-life assessment — Ancillary studies
  Other Names: quality of life assessment

SUMMARY:
This pilot clinical trial studies cryosurgery and radiation therapy in treating patients with painful bone metastases. Cryosurgery kills tumor cells by freezing them. Radiation therapy uses high-energy x-rays and other types of radiation to kill tumor cells and shrink tumors. Giving cryosurgery together with radiation therapy may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the potential for efficacy and safety of combining percutaneous computed tomography (CT)-guided cryoablation and radiotherapy for the palliation of osseous metastases.

OUTLINE:

Patients undergo cryosurgery. Beginning 2 weeks later, patients undergo 1, 10, or 15 fractions of radiation therapy 5 days per week for 1-3 weeks. Treatment continues in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 24 hours and weeks 1-2, 4, 12, 18, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Pathologically (histologically or cytologically) confirmed metastatic disease with a new tumor involving or abutting bone that has the clinical and imaging features of metastatic disease

  * If the nature of the metastatic disease has been previously documented, index tumor to be treated does not require further documentation (i.e., biopsy)
* Current analgesic therapies have failed (worst pain of 4 or above as measured by Brief Pain Inventory [BPI], despite analgesic therapy) OR the subject is experiencing intolerable side effects that preclude analgesic use (resulting in pain of 4 or above, as measured by BPI)
* Pain must be from one or two painful metastatic sites in the bone (additional less painful metastatic sites may be present)

  * Pain from the reported one or two metastatic sites must correlate with an identifiable tumor on CT, magnetic resonance imaging (MRI), or ultrasound (US) imaging
  * Metastatic tumors must be amenable to cryoablation with CT or MRI
* If the index tumor is in the spine, there must be an intact cortex between the mass and the spinal canal and exiting nerve roots
* Patients must have stable use of hormonal therapy for two weeks prior to study registration and two weeks prior to cryoablation procedure)
* Stable use of pain medications (no changes within two weeks of cryoablation procedure)
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* Life expectancy >= 2 months
* Platelets > 50,000/mm^3
* International normalized ratio (INR) >= 1.5
* Patients may not have any debilitating medical or psychiatric illness that would preclude giving informed consent or receiving optimal treatment and follow-up
* Patients who are taking antiplatelet or anticoagulation medication (e.g., aspirin, ibuprofen, low molecular weight heparin [LMWH] preparations) must be able to discontinue such treatment prior to the cryoablation procedure for an appropriate amount of time; at least 5 days should be allowed after discontinuation of aspirin, Coumadin, clopidogrel, and dipyridamole; at least 12 hours should be allowed after discontinuation of LMWH preparations
* Patients must be clinically suitable for cryoablation therapy
* Patients must be clinically suitable for radiation therapy
* Patients must be able to understand and willing to sign a written informed consent document

Exclusion Criteria:

* Patients with a diagnosis of leukemia, lymphoma, or myeloma
* Patients with a tumor involving a weight-bearing long bone of the lower extremity with the tumor causing > 50% loss of cortical bone
* Patients who have undergone prior ablation treatment or radiation therapy of the index tumor
* Patients who have received chemotherapy within 14 days prior to and 14 days after cryoablation procedure
* Index tumor(s) causing clinical or radiographic evidence of spinal cord or cauda equine compression/effacement
* Anticipated treatment of the index tumor that would require iceball formation within 1.0 cm of the spinal cord, brain, other critical nerve structure, large abdominal vessel such as the aorta or inferior vena cava (IVC), bowel, or bladder
* Any prior surgery at the proposed treatment site OR any prior surgery involving the cryoablation-treated tumor
* Index tumor involves the skull (treatment of other painful tumors in subjects with skull tumors is not excluded)
* Patients with uncontrolled coagulopathy or bleeding disorders
* Patients who are pregnant, nursing, or who wish to become pregnant during the study
* Patients with active, uncontrolled infection
* Patients with serious medical illnesses, including any of the following: uncontrolled congestive heart failure, uncontrolled angina, myocardial infarction, cerebrovascular event within six months prior to study entry
* Patients who are concurrently participating in any other experimental studies that could affect the primary endpoint of this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Childs, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Pain Level at 24 Hours Before Cryosurgery, as Measured by the BPI
Description: Numerical scores (0-10) from the BPI will be used to measure pain levels. Higher scores denotes worse outcome.
Time Frame: 24 hours
Measure: Number; unit: score on a scale
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
Number analyzed (Participants) | 1
score on a scale | 5

2. Secondary Outcome: Pain Medication Level, Assessed by Changes in Narcotic Medication Usage
Description: Pain medication assessments will be used to quantify any change in narcotic medication usage using the 24-hour morphine equivalent dose.
Time Frame: Baseline to 24 weeks
Measure: Number; unit: mg
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
Number analyzed (Participants) | 1
mg | 2

3. Secondary Outcome: Adverse Events, Graded According to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0
Time Frame: Up to 24 weeks
Measure: Number; unit: events
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
Number analyzed (Participants) | 1
events | 0

4. Secondary Outcome: Pain After Cryosurgery, as Measured by the BPI
Description: Questions #4 (least pain), #5 (average pain), and #6 (right now) from the BPI (reported on 0-10 scale) will be used as the secondary outcome measures. Higher scores denotes worse outcome
Time Frame: Up to 24 weeks
Measure: Number; unit: score on a scale
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
Number analyzed (Participants) | 1
score on a scale
  Least pain | 7
  Average Pain | 10
  Right now | 2

5. Secondary Outcome: Number of Participants Who Survived
Description: Count of participants that survived.
Time Frame: Up to 24 weeks post-cryosurgery
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
Number analyzed (Participants) | 1
Participants | 1

ADVERSE EVENTS:
Arm/Group | Treatment (Cryosurgery and Radiation Therapy)
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes